CLINICAL TRIAL: NCT05984394
Title: Evaluation of Antigen-specific Th1 and T17 Cells, ILC and MAIT in Patients With Antisynthetase Syndrome and Interstitial Lung Disease
Brief Title: Evaluation of Antigen-specific T Cells in Patients With Antisynthetase Syndrome and Interstitial Lung Disease
Acronym: CYTILDASS
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Paul DECKER, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023-A00804-41
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Antisynthetase Syndrome
MeSH Terms: conditions — Antisynthetase syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AS patients with ILD: New diagnosis of patients with AS syndrome and ILD
  Interventions: Diagnostic Test: BAL antigen-specific Th1 cells and Th17 cells, ILC and MAIT

INTERVENTIONS:
Diagnostic Test: BAL antigen-specific Th1 cells and Th17 cells, ILC and MAIT — BAL antigen-specific Th1 cells and Th17 cells, ILC and MAIT

SUMMARY:
Antisynthetase syndrome (AS) is a rare overlapping myositis characterized by cellular and humoral autoimmune responses directed against aminoacyl-tRNA synthetases. Intesrtitial lung disease (ILD) is a leading cause of mortality in antisynthetase syndrome. Recently, antigen-specific IFN-γ+ CD4+ T cells have been identified in bronchoalveolar fluid (BAL) of patients with antisynthetase syndrome and ILD. Elevated levels of IL1β, IL12, IL18, TNFα, IL17A, IL22 have also been detected in peripheral blood of AS patients, especially those with progressive ILD. Implication of innate lymphoid cells (ILC) and mucosal-associated invariant T cells (MAIT) have not yet been studied in patients with AS. Targeted therapies against Th1 and Th17 cells may represent a promising treatment in patients AS patients with ILD.

Investigators suppose that antigen-specific Th1 and Th17 cells, ILC and MAIT at ILD diagnosis are associated with ILD severity at diagnosis and could predict treatment response at 6 months.

The main objective is to study the correlation between BAL antigen-specific Th1 and Th17 cells at ILD diagnosis and clinical evolution after 6 months of treatment according to initial ILD severity.

ELIGIBILITY:
Inclusion Criteria:

* Patient with new diagnosis of AS with ILD

Exclusion Criteria:

* Patient with ILD differential diagnosis
* Corticosteroid treatment, immunosuppresive or immunomodulatory drugs in the past 3 months before diagnosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with AS and ILD
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
BAL antigen-specific Th1 and Th17 cells | baseline (J0)
  BAL antigen-specific Th1 and Th17 cells percentages among BAL total CD4+ T cells
FVC relative change | within 6 months after diagnosis
  Relative change of FVC percentage

SECONDARY OUTCOMES:
BAL antigen-specific Th1 and Th17 cells | baseline (J0)
  BAL antigen-specific Th1 and Th17 cells percentages among total BAL CD4+ T cells
FVC | baseline (J0)
  FVC percentage at ILD diagnosis
FVC absolute change | within 6 months after diagnosis
  Absolute change of FVC percentage
Global activity | baseline (J0)
  MDAAT score

OTHER OUTCOMES:
BAL ILC | baseline (J0)
  BAL ILC percentage among total BAL lymphoid cells
BAL MAIT | baseline (J0)
  BAL MAIT percentage among total BAL T cells

CONTACTS AND LOCATIONS:
Overall Officials: Paul Decker, MD, Principal Investigator — CHU NANCY
Locations (6):
- France (6):
  - Bernard Bonnotte, Dijon
  - Julien Campagne, Metz
  - Paul Decker, Nancy
  - Olivier Benveniste, Paris
  - Loïs Bolko, Reims
  - Alain Meyer, Strasbourg

IPD SHARING:
Plan to Share IPD: No